CLINICAL TRIAL: NCT06303336
Title: Effects of Neuromuscular Electrical Stimulation With and Without Dynamic Bracing on Lower Extremity Spasticity and Quality of Movement in Children With Cerebral Palsy
Brief Title: Effects OF NMES With and Without Dynamic Bracing on Spasticity and Movement Quality in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/0258 Ayesha Ashraf
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Diplegic Spastic Cerebral Palsy
Keywords: NMES; Dynamic Bracing; Cerebral Palsy; lower extremity
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participants and outcome assessors will be kept blind about the intervention which the patients will be receiving
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NMES with Dynamic Bracing (Experimental): The NMES targeting the hip adductors, the knee flexor muscles and the ankle & foot muscles, along with dynamic bracing
  Interventions: Other: NMES with Dynamic Bracing
- NMES without Dynamic Bracing (Experimental): Neuromuscular Electrical Stimulator targeting the lower extremity
  Interventions: Other: NMES without Dynamic Bracing
- Dynamic Bracing Only (Experimental): Dynamic Bracing of lower extremity
  Interventions: Other: Dynamic Bracing Only

INTERVENTIONS:
Other: NMES with Dynamic Bracing — The group will receive NMES along with dynamic bracing
  Arms: NMES with Dynamic Bracing
Other: NMES without Dynamic Bracing — The participants will receive NMES on the lower extremity
  Arms: NMES without Dynamic Bracing
Other: Dynamic Bracing Only — This group will receive dynamic bracing only on the lower limb.
  Arms: Dynamic Bracing Only

SUMMARY:
The study aims at comparing Neuromuscular electrical Stimulation with and without dynamic bracing on spasticity and movement quality of lower limb in Children with Cerebral Palsy

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a lifelong motor impairment caused by an early brain injury and affects 2-3 per 1,000 live births. It is a complex medical condition that negatively impacts cognition, language, sensations, movement, and gait patterns. It is normally carried out using a comprehensive approach that incorporates numerous approaches targeted at minimizing symptoms and improving functional outcomes.

NMES (Neuromuscular and Muscular Electrical Stimulation) is an instrument that provides electrical impulses to nerves, causing muscles to contract, while dynamic bracing use muscle power to pre-compress soft tissue to produce the high forces required to control specific pathological diseases.

The hip adductors, the knee flexor muscles, and the ankle and foot muscles (gastrocnemius and soleus may experience increased tone, causing the ankles to be held in a plantar-flexed (pointed downward) position) are targeted with NMES in the lower extremity to reduce the spasticity & improve the quality of movement in CP children. Investigating how combining NMES with dynamic bracing benefits lumbar disc bulge patients adds to the growing body of evidence supporting multimodal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 to 12 years.
* Able to walk with or without an assistive device. Classification as level I-II on the Gross Motor Functional Classification System (GMFCS).
* Able to stand with or without support for 1 minute.
* Classification as levels I-III on the Manual Ability Classification System (MACS); and the ability to follow and accept verbal instructions.
* Muscle tone scored ≥2, according to Modified Ashworth Scale.

Exclusion Criteria:

* Orthopedic Surgical intervention (e.g. tendon lengthening in lower limb) within the previous 12 months
* Treatment with botulinum toxin in the calf muscles within the previous 6 months
* Presence of structural deformities at the lower limbs and trunk, or instability in the ankle joint, which could compromise the child's safety and performance of the motor task
* Severe affective or psychiatric impairments;
* Serious vision or hearing problems
* Any neurological impairment (epilepsy or any other disease that would interfere with physical activity)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | baseline and 6 weeks
  The scale is used to measure spasticity minimum score is 0 and maximum score is 4
Observable Movement Quality Scale | baseline and 6 weeks
  it is used assess the movement quality in children Minimum Score: 0 (indicating the poorest movement quality) and maximum is 24
Physicians Rating Scale | baseline and 6 weeks
  it is used to objectively documenting the hip, knee, ankle and foot changes in children with CP. Minimum Score: 0 (indicating no impairment or lowest severity) and Maximum score is 7

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Ashraf, MS NMPT*, Principal Investigator — Ripha International Univerisity; Ammara Abbas, tDPT, Principal Investigator — Riphah International University
Locations (1):
- Children Hospital, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No